CLINICAL TRIAL: NCT05920317
Title: Retrospective Study of the Use of PRAEVAorta 2 Software for Vessel Geometric Analysis Versus Standard Analysis Methods in Patients With Abdominal Aortic Aneurysm
Brief Title: Comparison of a Full Automatic Software With Standard Methods of Vessels Analysis
Acronym: PRAEVA-2-LP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nurea (Industry)
Collaborators: Universitätsklinikum Leipzig (Other)
Responsible Party: Sponsor
Other Study IDs: PRAEVA-2-LP_CIP
Record Dates: First submitted 2022-03-02; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-05

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Aneurysm; AAA; software; Automatic; Scan
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Principal group: Analysis of the CT scans

SUMMARY:
The treatment of aortic aneurysms is today based on different indicators (diameters, lengths, angles, volumes of the arteries) measured on CT scan images. Several indicators are time consuming and complicatated to measure. They demand training and practice. Nurea is developing a software for automatic measurement of these indicators, PRAEVAorta® 2, to facilitate and assist the physician in his clinical routine.

The purpose of this study is to compare the analysis realised by the software PRAEVAorta® 2 with the analysis realised by the healthcare professional on retrospective CT scan images.

Contrasted and non-contrasted, pre-operation or post-operation CT scans from 50 patients will be analysed.

The main objectif is to validate the accuracy of the software by demonstrating its adequacy to the standard method of analysis.

The second objectives are the following:

* Evaluate the security of the software PRAEVAorta® 2
* Evaluate the unanticipated risks related to the use of the software
* Validate the accessory PRAEVAorta® Web

We make the following assumption :

90% of the patients show 90% of adequacy to the healthcare professional analysis

DETAILED DESCRIPTION:
The study PRAEVA-2-LP is realized in the University hospital of Leipzig. The treatment of aortic aneurysms is today based on different indicators (diameters, lengths, angles, volumes of the arteries) measured on CT scan images. Several indicators are time consuming and complicatated to measure. They demand training and practice. Nurea is developing a software for automatic measurement of these indicators, PRAEVAorta® 2, to facilitate and assist the physician in his clinical routine.

The purpose of this study is to compare the analysis realised by the software PRAEVAorta® 2 with the analysis realised by the healthcare professional on retrospective CT scan images.

Contrasted and non-contrasted, pre-operation or post-operation CT scans from 50 patients will be analysed.

We make the following assumption: 90% of the patients show 90% of adequacy to the healthcare professional analysis

This study is comparative, retrospective, non-interventional and monocentric. We compare the SaMD measurements to measurements realised using the standard method by a healthcare professional. The study analysis retrospective pseudonymised CT scans and deliver aggregated data. The study will be realised on a group of 50 subjects, which is small enough to have one site of investigation. Subjects will be their own witness. This strategy allows us to minimize the cost and the risks of the study without compromising the investigation. This investigation is submitted to the local ethics committee for approval according to paragraph 15 of Professional Code of the Saxon State Medical Association (Berufsordnung - BO) of 24 June 1998.

The study realised on the first version of the medical device PRAEVAorta® has shown a proportion of 93% of patient with measures calculated by the software in adequation with the measures realised following the standard method of analysis (ratio ≥ 90%). Because the new version of the software PRAEVAorta®2 has been improved, we expect to observe the same proportion.

Patient number calculation:

Hypotheses are the following:

H0: The proportion of patients with an absolute mean discrepancy > 5mm is 90% H1: The proportion of patient with an absolute mean discrepancy ≤ 5mm is strictly over 90% For this statistical analysis, variables are quantitative: aorta measurements. We consider over here the proportion of patients per sub-group who have as less or greater than 90%.

Comparison of two proportions: a theoretical proportion with an observed proportion The theoretical proportion ϕ0 is 90% The observed proportion ϕ is 93% (the observed proportion in the study of PRAEVAorta® 1) Therefore, the numbers of patients needed, with an α risk of 5% and a β risk of 0.9% is 32 in unilateral n=([1,96(φ0(1-φ0))^0,5 +u2β(φ(1-φ))^0,5]^2)/([φ0-φ]^2)=32 For security reasons and to anticipate any problem we choose to include approximately 10% more subjects. Moreover, to be sure that the amount of data is sufficient for CE marking we add another 15%. Therefore, the total of patient is 50.

The collected data comes from a database built by the hospital especially for retrospective study. The patient consent has already been collected at the creation of the database which exempt us from collecting it again.

The collected data are the gender, the birthdate of the patient, the scan manufacturer, the contrast-enhanced CT scan, the date of realization of the CT scan, the indicators, the healthcare professional trust in the results of the analysis realized by the software.

Images' analysis Pseudonymised images in DICOM format will be analysed. Pre-operation and post-operation thin-sliced CT images will be analysed.

Procedure to follow:

1. Inclusion and exclusion criteria validation
2. Demographic data and scanner references collection
3. CT scans (in DICOM format) collection
4. First Randomisation of the subjects' order
5. Determination of the measures by the physician with the standard method
6. Second randomisation of the subjects' order
7. Software analysis of the images with PRAEVAorta® 2 and Physician trust opinion In step 7, physicians will have to indicate if, based on the report generated by PRAEVAorta® 2, they trust the software measures or they do not, in order to validate clinical safety.

The comparison of data will be done during the statistical analysis.

The data will be collected in an EDC / e-CRF. The software allow authentication, account management with several level of access to the different parts and data. Exchanges are secured and data are stored on a Health Data Host accredited server. A back-up is regularly made.

The practician fills a form / report when measuring the indicators and the software PRAEVAorta® 2 is returning a pdf report. The data collected in the EDC will be compared with the data present in those two reports and in the hospital study database.

Most monitoring will be realised in remote. A monitoring visit will be realised at mid-time. A data review and validation will be realised before database lockdown. Data will then be validated by the PI and the data manager.

Data management:

Data collected are pseudonymised to ensure confidentiality and medical secret and registered in the e-CRF.

Demographic data as well as scans are available in the hospital's database, set up specifically for retrospective data studies. Measures realised on the CT scans are registered on an electronic report, for both measurements methods. The data from those reports and from the database are reported in the e-CRF. Analysed CT scans are also uploaded in the e-CRF.

Data cannot be registered in the software before the subject's inclusion has been validated.

Data entered into the software must be double-checked to limit errors.

Data validation:

This requirement is achieved through Source Data Verification, the process by which the information reported on the e-CRF by the investigator is compared with the original medical records to ensure it is complete and accurate during monitoring visits and closure visit.

In addition, a system of dynamic consistency checks is implemented in the e-CRF for rapid data validation when applicable.

Through the Source Data Validation process, the monitor should confirm accurate transcription of data from source files to the CRF and that the CRF contains all the relevant information about the patient's participation in the clinical trial.

Monitoring visit process

Process:

The first monitoring visit will be conducted after the completion of the Step 4. of the procedure has been completed, to review first part of data. The rest will be reviewed in close-out visit.

Monitoring call and conference will be realized at the end of each step and when required The Monitoring visit will review all of the responsibilities listed above. Following each monitoring visit / call, a monitoring report will be submitted to the QI.

The following activities may take place during each monitoring visit:

The following participant data will be source data verified for the indicated percentage of participants enrolled in the trial and all incidences reported since the last monitoring visit:

100% of eligibility criteria 100% of participant CRFs

Any updates and/or revisions to the following study documents since the last monitoring visit will also be reviewed:

Training documentation/records and Task Delegation Log updates Regulatory documentation including Health Canada approval/amendments

The following activities may be conducted at each monitoring visit:

Trial Master File

* Ensure that essential document files are complete and current.

Investigator and Site Personnel Responsibilities

* Ensure that the Task Delegation Log is complete and signed.
* Verify that the QI and site personnel are adhering to the protocol and conducting the study according to regulatory requirements, Procedures and NF ISO 14155:2020.
* Verify that study activities are being performed by the QI or have been delegated to personnel qualified by appropriate education and training.
* Provide and document any necessary training for the QI and site personnel, such as training on NF ISO 14155:2020, procedures, protocol, e-CRF…

CRF Review / Source Documentation Verification. Verify the following:

* Accurate, complete, and current source documentation is maintained.
* Participants' eligibility reviewed and signed off by QI/Sub-Investigator.
* All procedures outlined in the protocol were completed.
* Protocol deviations documented and reported according to the protocol.
* All dropouts of enrolled subjects are recorded in the source documentation and on the CRF.
* The QI has reviewed, signed, and dated all required e-CRF pages in a timely manner
* Data entries in the e-CRF pages coincide with the source documentation, and note any errors, omissions, or discrepancies by issuing queries within the e-CRF system and revise other bullets.
* Provide the site staff with copies of Data correction forms.
* Verify that previously outstanding data queries have been resolved, signed, and dated by the QI or designee.

Device Deficiency (DD)

* Verify all newly reported DDs against source documentation.
* Follow up on previously reported DDs
* Confirm that all DDs have been reported to the Sponsor
* Identify any unreported DDs in source documentation.
* Review DDs reporting procedures, as necessary.

Protocol Deviations

* Verify that all protocol deviations are documented appropriately in each participant's research record and on the appropriate protocol deviation form.
* Ensure that the site has reported all protocol deviations to the Ethical Committee, as defined by EC policy and/or procedures
* Address any protocol deviations with site personnel during the monitoring visit and identify ways to prevent a recurrence of similar issues.

General

* Confirm all data is verifiable against source documentation.
* Confirm no transcription errors have been made.
* Ensure corrections are lined out, dated & initialed (no erasures or "whiteouts").

Visit Conclusion

At the conclusion of the visit, the monitor will meet with the QI and site research staff to review visit findings and answer questions. The monitor will discuss the following topics at a minimum:

* Enrolment progress.
* Study conducts and documentation of study activities.
* Deviations.
* Scheduling of the next Monitoring Visit when applicable

Statistics:

Aggregated data analysed as treated and per subgroup. Descriptive analysis

* Pearson's coefficient correlation
* Absolute mean discrepancy per measurements
* Global mean and standard deviation per measurement endpoint
* Ratio for a measure
* Maximum aortic diameter ratio
* Computational analysis time The duration of the semi-automatic segmentation manually corrected by the 2 surgeons was reported and compared to the fully automatic method.
* Detectable and non-detectable error rate for safety evaluation
* Calculation of false positive, false negative, sensibility, specificity, positive predictive values, negative predictive values and likelihood ratio (LR+ and LR-).

Inferential analysis Objective: comparing an observed proportion p1 with a theoretical proportion p0 p1: proportion of adequate data p0: theoretical proportion: 90%

A one-sided right test will be realised to evaluate the comparison

Evaluation criteria:

Principal criteria:

* 90% of the patients shaw 90% of adequacy.

Secondary criteria:

Evaluation of the measurements and the segmentations:

* The mean discrepancy shall be ≤ 5mm
* Pearson correlation shall be ≥ 90%

Evaluation of risks:

* Unanticipated risks should not be critical Evaluation of the security
* The detectable error rate shall be ≥ 95%
* The non-detectable error rate shall be ≤ 5% Evaluation of PRAEVAorta® Web
* No critical bug No critical unanticipated risks

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients diagnosed with an infrarenal AAA and treated with EVAR at the University Hospital of Leipzig between 2015-2021
* Patient equal to or over 18 years old

Exclusion Criteria:

Patients with

* para-renal or thoraco-abdominal aortic aneurysms,
* associated iliac artery aneurysms,
* ruptured aneurysms,
* aortic dissections,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with diagnosed or suspicion of an abdominal aortic aneurysm.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-11-28 (Estimated); Study Completion 2023-12-28 (Estimated)

PRIMARY OUTCOMES:
Orthogonal maximum diameter of the aorta (mm) | 3 months
Thoraco-Aortic lengths of the aorta (mm) | 3 months
  * Proximal neck length
  * Infrarenal Aortic length
  * Left common Iliac artery length
  * Right common Iliac artery length
Infrarenal volume of the aorta (cm3) | 3 months
  * Volume circulating
  * Intraluminal thrombus volume
  * Total volume
Aorta and iliacs diameters at several places (mm) | 3 months
  * Aortic diameter above the uppermost renal artery
  * Upper proximal Neck Diameter
  * Neck Diameter 5mm under the lower renal
  * Neck Diameter 10mm under the lower renal
  * Neck Diameter 15mm under the lower renal
  * Neck diameter 20mm under the lower renal
  * Lower proximal Neck Diameter
  * Proximal right common Iliac artery Diameter
  * Middle right common iliac artery Diameter
  * Distal right common Iliac artery Diameter
  * Distal right external iliac artery Diameter
  * Proximal left common Iliac artery Diameter
  * Middle left common iliac artery Diameter
  * Distal left common iliac artery Diameter
  * Distal left external Iliac Diameter
  * Aortic bifurcation diameter
Suprarenal angulation (in degree) | 3 months
  Angle between the suprarenal aorta and the neck
Infrarenal angulation (in degree) | 3 months
  Angle between the neck and aneurysm

SECONDARY OUTCOMES:
Healthcare professional trust questionnaire | 2 days
  Do the professional trust or not the result returned by the software ? Yes or No reported in the CRF
Scan analyse time from segmentation to measurements | 3 months
  Time for analysis by the surgeon from segmentation to measurements Time for analysis by the automatique software from segmentation to measurement
Unanticipated risks | 3 days
  Risks that haven't been anticipated by Nurea, related to the use of the software
Number of male and female | 1 day
  the patient sex is collected in the CRF
Number of patient per age | 1 day
  the patient age is collected in the CRF

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Dr. Med. BRANZAN, Principal Investigator — UNIVERSITY CLINIC LEIPZIG AöR
Locations (1):
- Universitätsklinikum leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moll FL, Powell JT, Fraedrich G, Verzini F, Haulon S, Waltham M, van Herwaarden JA, Holt PJ, van Keulen JW, Rantner B, Schlosser FJ, Setacci F, Ricco JB; European Society for Vascular Surgery. Management of abdominal aortic aneurysms clinical practice guidelines of the European society for vascular surgery. Eur J Vasc Endovasc Surg. 2011 Jan;41 Suppl 1:S1-S58. doi: 10.1016/j.ejvs.2010.09.011. No abstract available. PMID 21215940
- [Background] Szilagyi DE, Elliott JP, Smith RF. Clinical fate of the patient with asymptomatic abdominal aortic aneurysm and unfit for surgical treatment. Arch Surg. 1972 Apr;104(4):600-6. doi: 10.1001/archsurg.1972.04180040214036. No abstract available. PMID 5013802
- [Background] Scott RA, Wilson NM, Ashton HA, Kay DN. Influence of screening on the incidence of ruptured abdominal aortic aneurysm: 5-year results of a randomized controlled study. Br J Surg. 1995 Aug;82(8):1066-70. doi: 10.1002/bjs.1800820821. PMID 7648155
- [Background] Ashton HA, Buxton MJ, Day NE, Kim LG, Marteau TM, Scott RA, Thompson SG, Walker NM; Multicentre Aneurysm Screening Study Group. The Multicentre Aneurysm Screening Study (MASS) into the effect of abdominal aortic aneurysm screening on mortality in men: a randomised controlled trial. Lancet. 2002 Nov 16;360(9345):1531-9. doi: 10.1016/s0140-6736(02)11522-4. PMID 12443589
- [Background] Norman PE, Jamrozik K, Lawrence-Brown MM, Le MT, Spencer CA, Tuohy RJ, Parsons RW, Dickinson JA. Population based randomised controlled trial on impact of screening on mortality from abdominal aortic aneurysm. BMJ. 2004 Nov 27;329(7477):1259. doi: 10.1136/bmj.38272.478438.55. Epub 2004 Nov 15. PMID 15545293
- [Background] Powell JT, Brown LC, Forbes JF, Fowkes FG, Greenhalgh RM, Ruckley CV, Thompson SG. Final 12-year follow-up of surgery versus surveillance in the UK Small Aneurysm Trial. Br J Surg. 2007 Jun;94(6):702-8. doi: 10.1002/bjs.5778. PMID 17514693
- [Background] Lederle FA, Johnson GR, Wilson SE, Chute EP, Littooy FN, Bandyk D, Krupski WC, Barone GW, Acher CW, Ballard DJ. Prevalence and associations of abdominal aortic aneurysm detected through screening. Aneurysm Detection and Management (ADAM) Veterans Affairs Cooperative Study Group. Ann Intern Med. 1997 Mar 15;126(6):441-9. doi: 10.7326/0003-4819-126-6-199703150-00004. PMID 9072929
- [Background] Walker TG, Kalva SP, Yeddula K, Wicky S, Kundu S, Drescher P, d'Othee BJ, Rose SC, Cardella JF; Society of Interventional Radiology Standards of Practice Committee; Interventional Radiological Society of Europe; Canadian Interventional Radiology Association. Clinical practice guidelines for endovascular abdominal aortic aneurysm repair: written by the Standards of Practice Committee for the Society of Interventional Radiology and endorsed by the Cardiovascular and Interventional Radiological Society of Europe and the Canadian Interventional Radiology Association. J Vasc Interv Radiol. 2010 Nov;21(11):1632-55. doi: 10.1016/j.jvir.2010.07.008. Epub 2010 Sep 29. No abstract available. PMID 20884242
- [Background] Ghouri M, Krajcer Z. Endoluminal abdominal aortic aneurysm repair: the latest advances in prevention of distal endograft migration and type 1 endoleak. Tex Heart Inst J. 2010;37(1):19-24. PMID 20200623
- [Background] Tonnessen BH, Sternbergh WC 3rd, Money SR. Mid- and long-term device migration after endovascular abdominal aortic aneurysm repair: a comparison of AneuRx and Zenith endografts. J Vasc Surg. 2005 Sep;42(3):392-400; discussion 400-1. doi: 10.1016/j.jvs.2005.05.040. PMID 16171578
- [Background] Wyss TR, Brown LC, Powell JT, Greenhalgh RM. Rate and predictability of graft rupture after endovascular and open abdominal aortic aneurysm repair: data from the EVAR Trials. Ann Surg. 2010 Nov;252(5):805-12. doi: 10.1097/SLA.0b013e3181fcb44a. PMID 21037436
- [Background] Vorp DA, Vande Geest JP. Biomechanical determinants of abdominal aortic aneurysm rupture. Arterioscler Thromb Vasc Biol. 2005 Aug;25(8):1558-66. doi: 10.1161/01.ATV.0000174129.77391.55. PMID 16055757
- [Background] Nicholls SC, Gardner JB, Meissner MH, Johansen HK. Rupture in small abdominal aortic aneurysms. J Vasc Surg. 1998 Nov;28(5):884-8. doi: 10.1016/s0741-5214(98)70065-5. PMID 9808857
- [Background] Powell JT, Sweeting MJ, Brown LC, Gotensparre SM, Fowkes FG, Thompson SG. Systematic review and meta-analysis of growth rates of small abdominal aortic aneurysms. Br J Surg. 2011 May;98(5):609-18. doi: 10.1002/bjs.7465. Epub 2011 Mar 17. PMID 21412998
- [Background] Lindholt JS, Vammen S, Juul S, Henneberg EW, Fasting H. The validity of ultrasonographic scanning as screening method for abdominal aortic aneurysm. Eur J Vasc Endovasc Surg. 1999 Jun;17(6):472-5. doi: 10.1053/ejvs.1999.0835. PMID 10375481
- [Background] Long A, Rouet L, Lindholt JS, Allaire E. Measuring the maximum diameter of native abdominal aortic aneurysms: review and critical analysis. Eur J Vasc Endovasc Surg. 2012 May;43(5):515-24. doi: 10.1016/j.ejvs.2012.01.018. Epub 2012 Feb 14. PMID 22336051
- [Background] Ellis M, Powell JT, Greenhalgh RM. Limitations of ultrasonography in surveillance of small abdominal aortic aneurysms. Br J Surg. 1991 May;78(5):614-6. doi: 10.1002/bjs.1800780529. PMID 2059819
- [Background] Leskinen R, Taskinen E, Volin L, Tukiainen P, Ruutu T, Hayry P. Use of bronchoalveolar lavage cytology and determination of protein contents in pulmonary complications of bone marrow transplant recipients. Bone Marrow Transplant. 1990 Apr;5(4):241-5. PMID 2159819
- [Background] Beales L, Wolstenhulme S, Evans JA, West R, Scott DJ. Reproducibility of ultrasound measurement of the abdominal aorta. Br J Surg. 2011 Nov;98(11):1517-25. doi: 10.1002/bjs.7628. Epub 2011 Aug 22. PMID 21861264
- [Background] Parr A, Jayaratne C, Buttner P, Golledge J. Comparison of volume and diameter measurement in assessing small abdominal aortic aneurysm expansion examined using computed tomographic angiography. Eur J Radiol. 2011 Jul;79(1):42-7. doi: 10.1016/j.ejrad.2009.12.018. Epub 2010 Jan 12. PMID 20061105
- [Background] Parr A, McCann M, Bradshaw B, Shahzad A, Buttner P, Golledge J. Thrombus volume is associated with cardiovascular events and aneurysm growth in patients who have abdominal aortic aneurysms. J Vasc Surg. 2011 Jan;53(1):28-35. doi: 10.1016/j.jvs.2010.08.013. PMID 20934838
- [Background] Stenbaek J, Kalin B, Swedenborg J. Growth of thrombus may be a better predictor of rupture than diameter in patients with abdominal aortic aneurysms. Eur J Vasc Endovasc Surg. 2000 Nov;20(5):466-9. doi: 10.1053/ejvs.2000.1217. PMID 11112467
- [Background] Houard X, Ollivier V, Louedec L, Michel JB, Back M. Differential inflammatory activity across human abdominal aortic aneurysms reveals neutrophil-derived leukotriene B4 as a major chemotactic factor released from the intraluminal thrombus. FASEB J. 2009 May;23(5):1376-83. doi: 10.1096/fj.08-116202. Epub 2009 Jan 9. PMID 19136615
- [Background] Houard X, Rouzet F, Touat Z, Philippe M, Dominguez M, Fontaine V, Sarda-Mantel L, Meulemans A, Le Guludec D, Meilhac O, Michel JB. Topology of the fibrinolytic system within the mural thrombus of human abdominal aortic aneurysms. J Pathol. 2007 May;212(1):20-8. doi: 10.1002/path.2148. PMID 17352452
- [Background] Satta J, Laara E, Juvonen T. Intraluminal thrombus predicts rupture of an abdominal aortic aneurysm. J Vasc Surg. 1996 Apr;23(4):737-9. doi: 10.1016/s0741-5214(96)80062-0. No abstract available. PMID 8627917
- [Background] Speelman L, Schurink GW, Bosboom EM, Buth J, Breeuwer M, van de Vosse FN, Jacobs MH. The mechanical role of thrombus on the growth rate of an abdominal aortic aneurysm. J Vasc Surg. 2010 Jan;51(1):19-26. doi: 10.1016/j.jvs.2009.08.075. Epub 2009 Nov 27. PMID 19944551
- [Background] Georgakarakos E, Ioannou CV, Kamarianakis Y, Papaharilaou Y, Kostas T, Manousaki E, Katsamouris AN. The role of geometric parameters in the prediction of abdominal aortic aneurysm wall stress. Eur J Vasc Endovasc Surg. 2010 Jan;39(1):42-8. doi: 10.1016/j.ejvs.2009.09.026. Epub 2009 Nov 10. PMID 19906549
- [Background] Kauffmann C, Tang A, Therasse E, Giroux MF, Elkouri S, Melanson P, Melanson B, Oliva VL, Soulez G. Measurements and detection of abdominal aortic aneurysm growth: Accuracy and reproducibility of a segmentation software. Eur J Radiol. 2012 Aug;81(8):1688-94. doi: 10.1016/j.ejrad.2011.04.044. Epub 2011 May 20. PMID 21601403
- [Background] Chaikof EL, Dalman RL, Eskandari MK, Jackson BM, Lee WA, Mansour MA, Mastracci TM, Mell M, Murad MH, Nguyen LL, Oderich GS, Patel MS, Schermerhorn ML, Starnes BW. The Society for Vascular Surgery practice guidelines on the care of patients with an abdominal aortic aneurysm. J Vasc Surg. 2018 Jan;67(1):2-77.e2. doi: 10.1016/j.jvs.2017.10.044. PMID 29268916
- [Background] Riambau V, Bockler D, Brunkwall J, Cao P, Chiesa R, Coppi G, Czerny M, Fraedrich G, Haulon S, Jacobs MJ, Lachat ML, Moll FL, Setacci C, Taylor PR, Thompson M, Trimarchi S, Verhagen HJ, Verhoeven EL, Esvs Guidelines Committee, Kolh P, de Borst GJ, Chakfe N, Debus ES, Hinchliffe RJ, Kakkos S, Koncar I, Lindholt JS, Vega de Ceniga M, Vermassen F, Verzini F, Document Reviewers, Kolh P, Black JH 3rd, Busund R, Bjorck M, Dake M, Dick F, Eggebrecht H, Evangelista A, Grabenwoger M, Milner R, Naylor AR, Ricco JB, Rousseau H, Schmidli J. Editor's Choice - Management of Descending Thoracic Aorta Diseases: Clinical Practice Guidelines of the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2017 Jan;53(1):4-52. doi: 10.1016/j.ejvs.2016.06.005. No abstract available. PMID 28081802
- [Background] Scott SW, Batchelder AJ, Kirkbride D, Naylor AR, Thompson JP. Late Survival in Nonoperated Patients with Infrarenal Abdominal Aortic Aneurysm. Eur J Vasc Endovasc Surg. 2016 Oct;52(4):444-449. doi: 10.1016/j.ejvs.2016.05.008. Epub 2016 Jun 30. PMID 27374814
- [Background] Claridge R, Arnold S, Morrison N, van Rij AM. Measuring abdominal aortic diameters in routine abdominal computed tomography scans and implications for abdominal aortic aneurysm screening. J Vasc Surg. 2017 Jun;65(6):1637-1642. doi: 10.1016/j.jvs.2016.11.044. Epub 2017 Feb 16. PMID 28216357
- [Background] Mell MW, Hlatky MA, Shreibati JB, Dalman RL, Baker LC. Late diagnosis of abdominal aortic aneurysms substantiates underutilization of abdominal aortic aneurysm screening for Medicare beneficiaries. J Vasc Surg. 2013 Jun;57(6):1519-23, 1523.e1. doi: 10.1016/j.jvs.2012.12.034. Epub 2013 Feb 12. PMID 23414696
- [Background] de Bruijne M, van Ginneken B, Viergever MA, Niessen WJ. Interactive segmentation of abdominal aortic aneurysms in CTA images. Med Image Anal. 2004 Jun;8(2):127-38. doi: 10.1016/j.media.2004.01.001. PMID 15063862
- [Background] Lopez-Linares K, Aranjuelo N, Kabongo L, Maclair G, Lete N, Ceresa M, Garcia-Familiar A, Macia I, Gonzalez Ballester MA. Fully automatic detection and segmentation of abdominal aortic thrombus in post-operative CTA images using Deep Convolutional Neural Networks. Med Image Anal. 2018 May;46:202-214. doi: 10.1016/j.media.2018.03.010. Epub 2018 Mar 27. PMID 29609054
- [Background] Ahmed S, Zimmerman SL, Johnson PT, Lai H, Kawamoto S, Horton KM, Fishman EK. MDCT interpretation of the ascending aorta with semiautomated measurement software: improved reproducibility compared with manual techniques. J Cardiovasc Comput Tomogr. 2014 Mar-Apr;8(2):108-14. doi: 10.1016/j.jcct.2013.12.009. Epub 2014 Jan 11. PMID 24568947
- [Background] Singh K, Jacobsen BK, Solberg S, Bonaa KH, Kumar S, Bajic R, Arnesen E. Intra- and interobserver variability in the measurements of abdominal aortic and common iliac artery diameter with computed tomography. The Tromso study. Eur J Vasc Endovasc Surg. 2003 May;25(5):399-407. doi: 10.1053/ejvs.2002.1856. PMID 12713777
- [Background] Caradu C, Spampinato B, Vrancianu AM, Berard X, Ducasse E. Fully automatic volume segmentation of infrarenal abdominal aortic aneurysm computed tomography images with deep learning approaches versus physician controlled manual segmentation. J Vasc Surg. 2021 Jul;74(1):246-256.e6. doi: 10.1016/j.jvs.2020.11.036. Epub 2020 Dec 9. PMID 33309556
- [Background] Taha AA, Hanbury A. Metrics for evaluating 3D medical image segmentation: analysis, selection, and tool. BMC Med Imaging. 2015 Aug 12;15:29. doi: 10.1186/s12880-015-0068-x. PMID 26263899
- [Background] Jongkind V, Yeung KK, Akkersdijk GJ, Heidsieck D, Reitsma JB, Tangelder GJ, Wisselink W. Juxtarenal aortic aneurysm repair. J Vasc Surg. 2010 Sep;52(3):760-7. doi: 10.1016/j.jvs.2010.01.049. Epub 2010 Apr 10. PMID 20382492
- [Background] Wever JJ, Blankensteijn JD, Th M Mali WP, Eikelboom BC. Maximal aneurysm diameter follow-up is inadequate after endovascular abdominal aortic aneurysm repair. Eur J Vasc Endovasc Surg. 2000 Aug;20(2):177-82. doi: 10.1053/ejvs.1999.1051. PMID 10942691
- [Background] Kritpracha B, Beebe HG, Comerota AJ. Aortic diameter is an insensitive measurement of early aneurysm expansion after endografting. J Endovasc Ther. 2004 Apr;11(2):184-90. doi: 10.1583/03-976.1. PMID 15056034
- [Background] van Keulen JW, van Prehn J, Prokop M, Moll FL, van Herwaarden JA. Potential value of aneurysm sac volume measurements in addition to diameter measurements after endovascular aneurysm repair. J Endovasc Ther. 2009 Aug;16(4):506-13. doi: 10.1583/09-2690.1. PMID 19702341
- [Background] Bley TA, Chase PJ, Reeder SB, Francois CJ, Shinki K, Tefera G, Ranallo FN, Grist TM, Pozniak M. Endovascular abdominal aortic aneurysm repair: nonenhanced volumetric CT for follow-up. Radiology. 2009 Oct;253(1):253-62. doi: 10.1148/radiol.2531082093. Epub 2009 Jul 31. PMID 19703867
- [Background] Nambi P, Sengupta R, Krajcer Z, Muthupillai R, Strickman N, Cheong BY. Non-contrast computed tomography is comparable to contrast-enhanced computed tomography for aortic volume analysis after endovascular abdominal aortic aneurysm repair. Eur J Vasc Endovasc Surg. 2011 Apr;41(4):460-6. doi: 10.1016/j.ejvs.2010.11.027. Epub 2010 Dec 31. PMID 21195639
- [Background] Prinssen M, Verhoeven EL, Verhagen HJ, Blankensteijn JD. Decision-making in follow-up after endovascular aneurysm repair based on diameter and volume measurements: a blinded comparison. Eur J Vasc Endovasc Surg. 2003 Aug;26(2):184-7. doi: 10.1053/ejvs.2002.1892. PMID 12917836
- [Background] Wanhainen A, Verzini F, Van Herzeele I, Allaire E, Bown M, Cohnert T, Dick F, van Herwaarden J, Karkos C, Koelemay M, Kolbel T, Loftus I, Mani K, Melissano G, Powell J, Szeberin Z, Esvs Guidelines Committee, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Kakkos S, Koncar I, Kolh P, Lindholt JS, de Vega M, Vermassen F, Document Reviewers, Bjorck M, Cheng S, Dalman R, Davidovic L, Donas K, Earnshaw J, Eckstein HH, Golledge J, Haulon S, Mastracci T, Naylor R, Ricco JB, Verhagen H. Editor's Choice - European Society for Vascular Surgery (ESVS) 2019 Clinical Practice Guidelines on the Management of Abdominal Aorto-iliac Artery Aneurysms. Eur J Vasc Endovasc Surg. 2019 Jan;57(1):8-93. doi: 10.1016/j.ejvs.2018.09.020. Epub 2018 Dec 5. No abstract available. PMID 30528142